CLINICAL TRIAL: NCT01832909
Title: Macronutrient Absorption From Walnuts: The Measured Energy Value of Walnuts in the Human Diet
Brief Title: The Measured Energy Value of Walnuts in the Human Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: California Walnut Board (Other)
Responsible Party: Principal Investigator, David Baer, Research Physiologist, USDA Beltsville Human Nutrition Research Center
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: HS43
Record Dates: First submitted 2013-04-08; First posted 2013-04-16 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Metabolizable Energy of Walnuts
Keywords: metabolizable energy; walnuts; Atwater factors; energy value

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Walnut Diet first, then Control Diet (Experimental): Controlled diet with 1.5 oz/d of walnuts, followed by controlled diet without walnuts.
  Interventions: Other: Walnut Diet; Other: Control Diet
- Control Diet first, then Walnut Diet (Experimental): Controlled diet without almonds first (control), then controlled diet with 1.5 oz/d of almonds.
  Interventions: Other: Walnut Diet; Other: Control Diet

INTERVENTIONS:
Other: Walnut Diet — Controlled diet with 1.5 oz/d of walnuts.
Other: Control Diet — Controlled diet without walnuts.

SUMMARY:
The objective of this study is to measure the energy value of walnuts in the human diet and study molecular mechanisms that may help explain the beneficial health effects of walnuts. The hypothesis is that there will be less metabolizable energy in walnuts due to decreased fat digestibility.

DETAILED DESCRIPTION:
Previous studies have demonstrated that nut consumption imparts a variety of health benefits, including reduction of cardiovascular disease and improved satiety. The aim of this study is to determine the energy value of walnuts in the human diet and to probe mechanisms by which walnuts impart health benefits. The metabolizable energy value of walnuts will be calculated based on the chemical composition and energy content of the consumed diet and excreta. This will provide a better estimate of the energy value of walnuts than simply calculating energy value based on Atwater factors. In addition to determining the energy value of walnuts, we will evaluate the effects of walnut-rich diets on plasma phytonutrient levels and on gene expression changes to determine what protective mechanisms are activated by walnut consumption.

ELIGIBILITY:
Inclusion Criteria:

* Age 25 to 65 years at beginning of study
* Body mass index between 20 and 38 kg/m2
* Fasting glucose < 126 mg/dl
* Blood pressure < 160/100 (controlled with certain medications)
* Fasting total blood cholesterol < 280 mg/dl
* Fasting triglycerides < 300 mg/dl

Exclusion Criteria:

* Presence of kidney disease, liver disease, gout, hyperthyroidism, untreated or unstable hypothyroidism, certain cancers, gastrointestinal disease, pancreatic disease, other metabolic diseases, or malabsorption syndromes
* Women who have given birth during the previous 12 months
* Pregnant women or women who plan to become pregnant or become pregnant during the study
* Lactating women
* Type 2 diabetes requiring the use of oral antidiabetic agents or insulin
* History of bariatric or certain other surgeries related to weight control
* Smokers or other tobacco users (during 6 months prior to the start of the study)
* Antibiotic use during the intervention or for 3 weeks prior to any intervention period
* History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians, very low fat diets, high protein diets)
* Volunteers who have lost 10% of body weight within the last 12 months
* Known (self-reported) allergy or adverse reaction to walnuts or other nuts
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past 12 months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Metabolizable Energy | Each three weeks, up to 6 weeks
  Metabolizable energy content will be calculated according to the methods of Novotny et al. (2012). Fat, protein, and fiber digestibility will be calculated and the effect of walnuts on nutrient digestibility will be assessed.

SECONDARY OUTCOMES:
Gene expression | At the end of each 3-week intervention period
  Gene expression in whole blood will be evaluated through global gene expression using the Affymetrix platform. Changes in specific genes observed with global gene expression technology will be confirmed through reverse transcription polymerase chain reaction.
Biomarkers of oxidative stress/inflammation | End of each 3-week intervention period
  Analysis of markers such as oxidized-low density lipoprotein and inflammatory markers (C-reactive protein, interleukin-1, interleukin-6, tumor necrosis factor-alpha).
Measure of walnut nutrients and metabolites | End of each 3-week intervention period
  Blood and urine will be analyzed for appearance of walnut nutrients and their metabolites.

CONTACTS AND LOCATIONS:
Locations (1):
- USDA Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

REFERENCES:
- [Background] Novotny JA, Gebauer SK, Baer DJ. Discrepancy between the Atwater factor predicted and empirically measured energy values of almonds in human diets. Am J Clin Nutr. 2012 Aug;96(2):296-301. doi: 10.3945/ajcn.112.035782. Epub 2012 Jul 3. PMID 22760558
- [Derived] Holscher HD, Guetterman HM, Swanson KS, An R, Matthan NR, Lichtenstein AH, Novotny JA, Baer DJ. Walnut Consumption Alters the Gastrointestinal Microbiota, Microbially Derived Secondary Bile Acids, and Health Markers in Healthy Adults: A Randomized Controlled Trial. J Nutr. 2018 Jun 1;148(6):861-867. doi: 10.1093/jn/nxy004. PMID 29726951
- [Derived] Baer DJ, Gebauer SK, Novotny JA. Walnuts Consumed by Healthy Adults Provide Less Available Energy than Predicted by the Atwater Factors. J Nutr. 2016 Jan;146(1):9-13. doi: 10.3945/jn.115.217372. Epub 2015 Nov 18. PMID 26581681